CLINICAL TRIAL: NCT05014698
Title: IDEntification of New Predisposition Genes in Differentiated THYroid Cancer
Acronym: IDENTHY-K
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: end-of-study visit not completed within the protocol timeframe
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC19_0414
Record Dates: First submitted 2021-08-05; First posted 2021-08-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Differentiated Thyroid Cancer; Thyroid Cancer, Nonmedullary
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WGS (Experimental): at inclusion visit :
  - Blood collection for whole Genome sequencing will be performed
  At final visit :
  the results of the WGS will be delivered to patients
  Interventions: Genetic: WGS

INTERVENTIONS:
Genetic: WGS — Whole Genome sequencing

SUMMARY:
The purpose of this research is to find new predisposition genes for differentiated thyroid cancer (DTC).

DETAILED DESCRIPTION:
The purpose of this research is to find new predisposition genes for differentiated thyroid cancer (DTC). Therefore, in the absence of a BAP1 and DICER1 abnormality, we offer to sequence your whole genome (WGS) or partial genome (genotyping) for a previously unknown genetic abnormality.

Furthermore, the discovery of new genes would be a major medical advance that could contribute to the identification of new therapeutic targets.

This research will be conducted at the University Hospital of Nantes and the Hospital of Vendée and 95 people should participate.

ELIGIBILITY:
Inclusion Criteria:

* Probant subjects
* Minor or adult subject
* Adult subject or legal guardian for minor subjects agreeing to sign the study consent and biospecimen consent
* Subject with differentiated thyroid cancer without an identified causative mutation in the BAP1 and DICER 1 predisposition genes
* Patient affiliated to a valid social security plan

Relative subjects

* Adult subjects
* Subject agreeing to sign the study consent and the biocollection consent
* Subject with differentiated thyroid cancer or from a family with several cases of differentiated thyroid cancer without a causal mutation identified in the BAP1 and DICER 1 predisposition genes
* Patient affiliated to a social security plan

Exclusion Criteria:

* Subject refusing to participate
* Subjects with a causal mutation identified in the predisposition genes: BAP1 and DICER 1
* Subjects under guardianship, curatorship or safeguard of justice or not socially insured
* Subjects with another syndromic predisposition to thyroid cancer (Cowden, Werner, PAF)

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2026-01-13 (Actual); Study Completion 2026-01-13 (Actual)

PRIMARY OUTCOMES:
Type and Number of genetic variants associated with or causing the development of differentiated thyroid cancer | within 2 years
  To be achieved by a whole genome sequencing (WGS) approach in a familial analysis of patients with differentiated thyroid cancer. In addition, high-throughput genotyping of multiple individuals in each family will allow complementary detection of genomic regions that are shared only by affected subjects

SECONDARY OUTCOMES:
Number of phenotypes associated to genotypes of CDT | within 2 years
  By studying the association between the clinical characteristics of patients and the identified genetic variants
Analysis of birthplace/family origin information | within 2 years
  Definition of the spatial location of family forms of CDT and to identify possible founding effects

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Vendée Hospital, La Roche-sur-Yon
  - Nantes University Hospital, Nantes

IPD SHARING:
Plan to Share IPD: No